CLINICAL TRIAL: NCT03352141
Title: Non-Invasive Fat Reduction With Cryolipolysis for Jawline Contouring
Brief Title: Cryolipolysis for Jawline Contouring
Acronym: JAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA17-004
Record Dates: First submitted 2017-11-08; First posted 2017-11-24 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fat Reduction (Experimental): The treatments are designed to see if the fat can be reduced along the jawline with Cryolipolysis.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting machine will be used to perform the treatments.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of non-invasive reduction of subcutaneous fat along the jawline with Cryolipolysis.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Treatment area skin fold thickness > 1cm (measured by caliper).
* Sufficient treatment area requiring at least 2 cooling cycles.
* No weight change exceeding 5% of body weight in the preceding month.
* Agreement to maintain his/her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject has signed a written informed consent form.

Exclusion Criteria

* Excessive skin laxity in the treatment area for which reduction of subcutaneous fat may, in the opinion of the investigator, result in an unacceptable aesthetic result.
* Prominent platysmal bands at rest which may interfere with assessment of treatment area.
* Evidence of any cause of enlargement in the treatment area other than localized subcutaneous fat, such as swollen lymph nodes or ptotic submandibular glands.
* Significant enlargement on the anterior neck that may prevent the proper placement of the applicator e.g. enlarged thyroid glands.
* Treatment with dermal fillers, radiofrequency or laser procedures, or chemical peels in the treatment area (below the mandible) within the past 6 months.
* Botulinum toxin or other aesthetic drug injections within the treatment area in the past 6 months.
* History of facial nerve paresis or paralysis (such as Bell's palsy).
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) or implant in or adjacent to the area of intended treatment.
* History of prior neck surgery, or prior surgery in the area of intended treatment.
* Current infection in and adjacent to treatment area.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 6 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brandt, BSN, Study Director — Zeltiq Aesthetics
Locations (1):
- Pacific Derm, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CoolSculpting for Jawline Contouring: All enrolled participants will be treated with the Zeltiq CoolSculpting System in the jawline area. Each participant will have up to 2 treatments, treatments 6 weeks apart.
Period: Overall Study
Arm/Group | CoolSculpting for Jawline Contouring
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CoolSculpting for Jawline Contouring
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Am Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 0
  Native Hawaiian or Other Pac Islander | 0
  White | 13
  Other | 1
Region of Enrollment [Number; unit: participants]
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unanticipated Adverse Device Effects (UADE)
Description: This outcome measurement considered all unanticipated device- or procedure-related adverse effects.
Time Frame: Enrollment through study completion, an average of 6 months.
Population: All 15 enrolled subjects were evaluated by the study investigator for unanticipated adverse device effects throughout the duration of the study.
Measure: Number; unit: Participants with UADE reported
Arm/Group | CoolSculpting for Jawline Contouring
Number analyzed (Participants) | 15
Participants with UADE reported | 0

2. Primary Outcome: Number of Before and After Side-by-side Photograph Pairs Correctly Identified by At Least 2 of 3 Blinded, Independent Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment (baseline) and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which photographs will be presented will be randomized; for each subject placement of the baseline and pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as 75% correct identification of pre-treatment photos by 2 out of 3 reviewers.
Time Frame: Baseline through 12 weeks post second treatment.
Population: Fourteen (14) of the enrolled subjects were included in the analysis of efficacy. One (1) subject was excluded due to body weight outside the requirements of the protocol.
Measure: Number; unit: Number Photo Pairs Correctly Identified
Units Other Than Participants: Photograph Pairs
Arm/Group | CoolSculpting for Jawline Contouring
Number analyzed (Participants) | 14
Number analyzed (Photograph Pairs) | 14
Number Photo Pairs Correctly Identified | 8

3. Secondary Outcome: Change in Fat Layer in the Treated Jawline Area
Description: When compared to baseline ultrasound imaging, the change in fat layer thickness at the final post-treatment visit will be measured. Ultrasound measurements were obtained in 5 areas intended for treatment at the baseline visit. A template was created for identification of the locations for subsequent measurements using external landmarks (e.g. skin imperfections) as reference points. The Treatment Effect = Follow-Up Average Thickness - Baseline Average Thickness. A negative change reflects a decrease in the average thickness from the baseline visit to the follow-up visit, and a positive result reflects an increase.
Time Frame: Baseline and 12 weeks post-final treatment.
Population: Fourteen (14) subjects were included in the efficacy analysis; one (1) subject was excluded due to weight change outside of the requirements of the protocol.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Submental Ultrasound Measurement; Submandibular Ultrasound Measurement (LEFT); Submandibular Ultrasound Measurement (RIGHT); Jowl Ultrasound Measurement (LEFT); Jowl Ultrasound Measurement (RIGHT): Fourteen subjects were included in the efficacy analysis. One subject was excluded due to weight change outside the requirements of the protocol.
Arm/Group | Submental Ultrasound Measurement | Submandibular Ultrasound Measurement (LEFT) | Submandibular Ultrasound Measurement (RIGHT) | Jowl Ultrasound Measurement (LEFT) | Jowl Ultrasound Measurement (RIGHT)
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
cm | -0.14 (0.12) | -0.10 (0.11) | -0.10 (0.11) | -0.08 (0.07) | -0.03 (0.05)

4. Secondary Outcome: Overall Satisfaction With the Treatment
Description: Subject satisfaction with the CoolSculpting procedure will be assessed by a questionnaire administered at the 12-week post-final treatment follow-up visit. The questionnaire will consist of 5-point Likert questions with 1 = very dissatisfied; 2 = dissatisfied; 3 = not sure; 4 = satisfied and 5 = very satisfied. Positive responses (very satisfied and satisfied) will be reported.
Time Frame: 12-week post-final treatment follow-up visit
Population: Fourteen subjects were included in the efficacy analysis. One subject was excluded due to weight change outside the requirements of the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting for Jawline Contouring
Number analyzed (Participants) | 14
Participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment through the final 12-week post-final treatment follow-up visit, an average of 6 months.
Arm/Group | CoolSculpting for Jawline Contouring
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting for Jawline Contouring (N=15)
Prolonged bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Prolonged edema (Skin and subcutaneous tissue disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03352141/Prot_SAP_001.pdf